CLINICAL TRIAL: NCT06612671
Title: Prognostic Factors and Oncological Outcome Analysis of Retroperitoneal Sarcoma
Brief Title: Treatment Outcomes of Retroperitoneal Sarcoma
Status: Active, not recruiting | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CE23365A
Record Dates: First submitted 2023-09-09; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Retroperitoneal Sarcoma
Keywords: Retroperitoneal Sarcoma; Surgery; Radiotherapy
MeSH Terms: interventions — Radiation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: tumor wide excision — patients received properative or post-operative radiotherapy
  Other Names: Radiation

SUMMARY:
Investigators tried condult a retrospective study to analysis the prognostic factors and oncological outcome analysis of Retroperitoneal Sarcoma treated in our high volume medical center.

DETAILED DESCRIPTION:
Retroperitoneal Sarcoma (RPS) which is a rare disease which incidence is 1.79/100,000. The treatment is difficult to due to it anatomy position which often invade to multiple organs and cause the complete surgical resection to be very complex and difficult. It was known to sacrifice one side kidney will improve the resection rate. To this days, successful surgical resection was still the gold standard that provide most benefit in overall survival. To reach that goal, pre-operative radiotherapy was applied to RPS which intended to achieve similar effect in rectal cancer for the down staging effect and improved the respectability but with limited benefit. Herein, investigators conducted this study to find the best way to achieve successful surgical resection and prognostic factor analysis.

ELIGIBILITY:
Inclusion Criteria:

* the patient who have retroperitoneal maliganacy and receive complete tumor excision in our hospital

Exclusion Criteria:

* the patient did not receive complete tumor excision in our hospital
* the pathological report yielded not malignancy tumor

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patient who have retroperitoneal maliganacy and receive complete tumor excision in our hospital. The preoperative procedure including angiography or TAE, radiotherapy is allowed.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | The proportion of patients still alive at 1 year, 3 years, and 5 years after treatment.
  After treatment, patients will undergo long-term follow-up to record their survival status.

SECONDARY OUTCOMES:
Progression free survival | The rates of local recurrence, regional recurrence, or distant metastasis at 1 year, 3 years, and 5 years after treatment.
  Progression defined as local, regional, or distant metastasis

OTHER OUTCOMES:
The resectability of preoperative embolization | From the start of preoperative evaluations to the day of surgery, it typically spans 7 days.
  Preoperative embolization for assessing resectability combines radiology, angiography, and transcatheter arterial embolization (TAE). Initially, imaging techniques such as X-rays or CT scans are used to understand the characteristics of the lesions. Then, angiography is employed to observe the tumor's blood supply. Finally, TAE not only evaluates the vascular supply to the tumor but also helps reduce its size through embolization, enhancing resectability. The comprehensive results of these assessments contribute to developing a safe and effective surgical plan.
The value of eGFR in renal function | Period from date before surgery to the date one year after suregry
  eGFR is an important biomarker used to assess kidney function and monitor renal health. It represents the volume of blood filtered by the glomeruli per minute, typically expressed in milliliters per minute (mL/min). A venous blood sample will be collected and analyzed in the laboratory to determine the value.

CONTACTS AND LOCATIONS:
Overall Officials: Radiation-Oncology Department Liu, M.D., Principal Investigator — Department of Radiation-Oncology, Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
I would like to share after the paper publish.